CLINICAL TRIAL: NCT04951661
Title: The Feasibility & Effectiveness of Virtual Reality in Reducing Pain for Older Adults With Knee Osteoarthritis
Brief Title: Virtual Reality and Older Adult Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Nancy Baker, Chair of and Associate Professor in Department of Occupational Therapy, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001433
Record Dates: First submitted 2021-06-10; First posted 2021-07-07 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Virtual Reality; Pain; Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): Participants will be set up in the VR equipment. They will engage and follow along with a 10-20 minute guided meditation through the VR. The meditation program may include simulated movement, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Participants will be set up in the VR equipment. They will engage and follow along with a 10-20 minute guided meditation through the VR. The meditation program may include simulated movement, relaxing music, and the voice of a meditation guide. The research team member will supervise the session, ensuring safety of the subject is maintained.

SUMMARY:
At the Brigham and Women's Hospital (BWH) Pain Management Center (PMC), knee OA is one of the most common conditions causing older adults to experience chronic pain. At this site, the core treatments of education, physical activity, and weight management are addressed, and then both pharmacological and nonpharmacological treatment options are available for patients living with chronic pain. Pharmacological treatments, such as topical and oral nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen, steroidal and non-steroidal injections, and prescription medications are currently the most commonly used treatments for chronic pain, but are also associated with limited benefits and dangerous side effects, such as addiction. Clients can also opt for nonpharmacological pain treatments at the PMC, such as acupuncture, reiki, physical therapy, and yoga, which are currently being researched at the clinic as well. The critical gap addressed with this pilot study is the need for additional safe and feasible treatment options for the growing population of older adults with chronic knee OA, as there is limited existing research on the effects of nonpharmacological treatments on this population. While past studies at the PMC have looked at the physiological mechanisms involved with chronic knee OA and the older adult population, the site has had limited funding to research nonpharmacological treatments such as virtual reality. In fact, there is limited evidence in the literature on the effects of virtual reality in reducing pain specifically for the older adult population.

DETAILED DESCRIPTION:
Virtual reality has been shown to be feasible for a variety of populations, including young people with autism experiencing specific phobia, pediatric burn patients, and young adults. However, there is limited evidence on the feasibility of VR for treating pain for the older adult population. Preliminary studies demonstrate the feasibility and safe qualities of immersive VR as a treatment tool for older adults with cognitive and physical impairments. One study demonstrated that older adults reported no negative side effects and 76% of the group wanted to try VR again. Furthermore, preliminary evidence on the feasibility of use in the clinic in terms of the construct of time was demonstrated.

Another study found that young adults and older adults who engaged in an immersive spatial navigation VR environment reported similar experiences, demonstrating that older adults experienced acceptable adverse effects and reported enjoyment through the VR immersion. Further recent studies provide evidence on the attitudes and treatment acceptability of older adults with chronic musculoskeletal pain towards VR as a distraction therapy for chronic pain exacerbations. These researchers discovered that 73.4% of the participants found VR to be an acceptable way to manage pain, and 73.3% reported they would be willing to use it for their pain. Only 26% of the participants experienced side effects such as general discomfort or eyestrain. Additionally, the qualitative data in this study suggests greater ease of use with sufficient practice and a preference towards relaxation, meditation, or biofeedback simulations with realistic images.

Thirty percent of older adults in the United States report experiencing chronic pain, with 41% of this subset of the population experiencing chronic joint pain. Knee osteoarthritis (OA) affects 37% of individuals aged 60 years or older who participated in the National Health and Nutrition Examination. This condition typically involves pain, stiffness, reduced joint motion and muscle weakness, and chronic pain that can have profound effects on physical function, psychological parameters, and overall quality of life. In knee OA, cartilage in the knee is lost and there is failed repair of joint damage, as OA is a disease of the whole joint. There is also often a discrepancy between severity of symptoms and severity of knee OA, which may relate to pain sensitization, adaptation to chronic pain, or reduction in activity to avoid pain.

In Virtual Reality (VR) people experience a three-dimensional, computer-generated environment via a computer headset. There are several mechanisms through which VR has been shown to effectively reduce pain. For one, gate theory of attention proposes that VR reduces perception of pain by absorbing and diverting attention away from pain. Dr. Brennan Spiegel, director of Cedars-Sinai Health Services Research, reports that VR's ability to distract the brain allows the brain to relax. He states that this modality "triggers signals that release natural pain-killing opioids from the spinal cord, essentially closing the gate, blocking the pain". Therefore, VR distraction may be a useful tool for clinicians who work with clients experiencing a variety of pain-related conditions, such as chronic knee osteoarthritis.

This pilot study will build off of these preliminary studies by working from the basis that older adults generally enjoy their immersive VR experience and including some of the relevant key requirements for immersive environments such as individual briefing and user-friendly handling. There are still many questions that need to be answered about the feasibility of VR as a clinical tool and its effectiveness in decreasing chronic pain, specifically for older adults. Therefore, this pilot study will look more into these topic areas through a subset of the population of older adults with chronic pain.

Currently, there has been very little research that has examined the effect of VR on chronic pain, particularly for the older adult population. Knowledge on the effectiveness of VR for chronic pain for older adults is necessary to determine best methods to feasibly integrate VR into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over the age of 60 years old (no upper limit)
2. Diagnosis of chronic knee osteoarthritis with pain in at least one knee
3. English-speaking
4. Willing and able to visit the PMC campus to participate in the study

Exclusion Criteria:

1. Received steroid injection within 2 weeks of VR session
2. Unwilling to put on VR headset
3. Diagnosed seizure disorder
4. Cognitive impairment
5. Hearing/visual deficit
6. Active, contagious skin infection
7. Eye infections
8. Has a pacemaker or defibrillator
9. Has a hearing aid

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Pain Numerical Rating Scale [NRS] (Change) | pre-intervention, within 20 minutes after intervention, 24-48 hour follow-up after intervention
  Measures the intensity of pain on an 11-point scale, ranging from 0-10. 0 is no "pain", and 10 is "pain as bad as you can imagine".
Brief Pain Inventory-Short Form (Change) | pre-intervention, 24-48 hour follow-up after intervention
  Fifteen-item self-report questionnaire that measures participant's various levels of pain severity in the past 24 hours, and perception of the degree to which pain prevents participation in important daily activities (e.g. work, socialization) and enjoyment of life. Eight pain severity items are rated on a 11-point scale of 0 (no pain) to 10 (pain as bad as you can imagine). Seven pain interference items are rated on a 11-point scale of 0 (does not interfere) to 10 (completely interferes).
PROMIS Emotional Distress - Short Form (Change) | pre-intervention, 24-48 hour follow-up after intervention
  24-item self report questionnaire that measures how often participant experiences feelings related to depression, anxiety and anger in the past seven days. These questionnaires have been modified to ask about the past 24 hours. The questionnaire uses a 5-point Likert scale, from 1 (never) to 5 (always). This questionnaire will assess the participant's psychological state.
Positive and Negative Affect Scale [PANAS] (Change) | pre-intervention, within 20 minutes after intervention, 24-48 hour follow-up after intervention
  This ten-item self-report questionnaire measures the extent to which the participant felt various emotions right now. This questionnaire uses a 5-point Likert scale, from 1 (very slightly or not at all) to 5 (extremely). This questionnaire will assess the participant's psychological state at all three data collection points.
Patient Global Impression of Change [PGIC] (Change) | within 20 minutes after intervention, 24-48 hour follow-up after intervention
  1-item self-report questionnaire that measures subject's pain since the start of the study intervention using a 7-point Likert scale from 0 (very much improved) to 6 (very much worse). This questionnaire will determine if the subject found the VR intervention to be helpful in reducing their pain.
Pain Catastrophizing Scale [PCS] (Change) | pre-intervention, 24-48 hour follow-up after intervention
  Thirteen-item self-report questionnaire that collects data on the types of thoughts and feelings the participants have when in pain. The participants will be asked to rank the degree to which they have certain thoughts and feelings when they are in pain using a 5-point Likert scale, from 0 (not at all) to 4 (all the time).
Survey of Pain Attitudes - Brief [SOPA] | pre-intervention
  30-item self-report questionnaire that measures participant's perceptions of and attitudes towards their pain. The participants will be asked to rank how true each statement is for them using a 5-point Likert scale, from 0 (very untrue) to 4 (very true).

SECONDARY OUTCOMES:
Baseline Survey | pre-intervention
  Obtains demographics, medical history, perceptions/attitudes of pain, and experiences with VR. Perceptions and attitudes towards pain will be obtained using the Pain Catastrophizing Scale17 and the Survey of Pain Attitudes19.
Simulator Sickness Questionnaire [SSQ]21 | within 20 minutes after intervention
  List of sixteen symptoms which are commonly experienced by users of virtual reality systems. Participants rate the severity of these symptoms while using the VR system using a 4-point Likert scale from 1 (none) to 4 (severe). This questionnaire will monitor the extent of motion sickness in our participants.
User Engagement Scale [UES]22 | within 20 minutes after intervention
  Twelve-item self-report questionnaire that measures the participant's perception of how engaged they were with the experience using a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). This questionnaire will determine immersion into VR.
iGroup Presence Questionnaire (IPQ) | within 20 minutes after intervention
  Fourteen-item self-report questionnaire that measures participant's perception of presence in computer-made Virtual Environments using various 7-point Likert scales. This questionnaire will determine immersion into VR.
Meditation Experience Questionnaire (MEQ) | within 20 minutes after intervention
  Thirteen-item self-report questionnaire that asks subjects to rate the frequency of occurrence of various experiences, such as fatigue, pleasant/unpleasant thoughts, and thoughts about planning or memories, during meditation intervention to evaluate quality of meditation immersion. Uses 5-point Likert scale from 1 (never) to 5 (almost constantly).
Open Ended Questions | within 20 minutes after intervention
  People in VR group will also be asked a series of open-ended questions about their experiences with VR and the study. Their responses will be audio recorded and later transcribed. These files will be stored in a password protected file that only study personnel have access to.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Baker, Principal Investigator — Tufts University
Locations (1):
- Brigham & Women's Pain Management Center, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Appel L, Appel E, Bogler O, Wiseman M, Cohen L, Ein N, Abrams HB, Campos JL. Older Adults With Cognitive and/or Physical Impairments Can Benefit From Immersive Virtual Reality Experiences: A Feasibility Study. Front Med (Lausanne). 2020 Jan 15;6:329. doi: 10.3389/fmed.2019.00329. eCollection 2019. PMID 32010701
- [Background] Billups, E. (2019, September 30). Hijacking the brain: Scientists are using VR to treat chronic pain. Spectrum News NY1. https://www.ny1.com/nyc/all-boroughs/exploring-your-health/2019/09/23/hijacking-the-brain--scientists-are-using-vr-to-treat-chronic-pain
- [Background] Bjordal JM, Klovning A, Ljunggren AE, Slordal L. Short-term efficacy of pharmacotherapeutic interventions in osteoarthritic knee pain: A meta-analysis of randomised placebo-controlled trials. Eur J Pain. 2007 Feb;11(2):125-38. doi: 10.1016/j.ejpain.2006.02.013. Epub 2006 May 8. PMID 16682240
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Hoffman HG, Meyer WJ 3rd, Ramirez M, Roberts L, Seibel EJ, Atzori B, Sharar SR, Patterson DR. Feasibility of articulated arm mounted Oculus Rift Virtual Reality goggles for adjunctive pain control during occupational therapy in pediatric burn patients. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):397-401. doi: 10.1089/cyber.2014.0058. PMID 24892204
- [Background] Jones T, Moore T, Choo J. The Impact of Virtual Reality on Chronic Pain. PLoS One. 2016 Dec 20;11(12):e0167523. doi: 10.1371/journal.pone.0167523. eCollection 2016. PMID 27997539
- [Background] Kennedy, S., & Moran, M. (2010). Pharmacological treatment of osteoarthritis of the hip and knee. BCMJ, 52(8), 404-9. https://bcmj.org/articles/pharmacological-treatment-osteoarthritis-hip-and-knee
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Maskey M, Rodgers J, Grahame V, Glod M, Honey E, Kinnear J, Labus M, Milne J, Minos D, McConachie H, Parr JR. A Randomised Controlled Feasibility Trial of Immersive Virtual Reality Treatment with Cognitive Behaviour Therapy for Specific Phobias in Young People with Autism Spectrum Disorder. J Autism Dev Disord. 2019 May;49(5):1912-1927. doi: 10.1007/s10803-018-3861-x. PMID 30767156
- [Background] Mendoza T, Mayne T, Rublee D, Cleeland C. Reliability and validity of a modified Brief Pain Inventory short form in patients with osteoarthritis. Eur J Pain. 2006 May;10(4):353-61. doi: 10.1016/j.ejpain.2005.06.002. Epub 2005 Jul 26. PMID 16051509
- [Background] Nakad, L., & Rakel, B. (2019). (271) Attitudes of Older Adults with Chronic Musculoskeletal Pain towards Immersive Virtual Reality. The Journal of Pain, 20(4), S42. https://doi.org/10.1016/j.jpain.2019.01.193
- [Background] NIH Pain Consortium. (n.d.). Chronic pain in older adults. https://www.painconsortium.nih.gov/sites/default/files/aging_and_chronic_pain_infographic_508.pdf
- [Background] Sakhare AR, Yang V, Stradford J, Tsang I, Ravichandran R, Pa J. Cycling and Spatial Navigation in an Enriched, Immersive 3D Virtual Park Environment: A Feasibility Study in Younger and Older Adults. Front Aging Neurosci. 2019 Aug 16;11:218. doi: 10.3389/fnagi.2019.00218. eCollection 2019. PMID 31474851
- [Background] Sharma L. Osteoarthritis of the Knee. N Engl J Med. 2021 Jan 7;384(1):51-59. doi: 10.1056/NEJMcp1903768. No abstract available. PMID 33406330
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Derived] Sarkar TD, Edwards RR, Baker N. The feasibility and effectiveness of virtual reality meditation on reducing chronic pain for older adults with knee osteoarthritis. Pain Pract. 2022 Sep;22(7):631-641. doi: 10.1111/papr.13144. Epub 2022 Jul 4. PMID 35750655